CLINICAL TRIAL: NCT03196271
Title: Evaluating the Tolerance, Compliance, Acceptability and Safety of Ketocal 2.5:1 LQ, a Nutritionally Complete Liquid Feed for Use as Part of the Ketogenic Diet (KD) in Children 8+ Years, Adolescents and Adults With Intractable Epilepsy or Other Disorders Where the KD is Indicated
Brief Title: Ketogenic Diet Drink Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K251 Study
Record Dates: First submitted 2017-05-26; First posted 2017-06-22 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Intractable Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Other): One single arm, consisting of a 3 day baseline period, a 28 day control period and a 28 day intervention period (Ketocal 2.5:1), in that order.
  Interventions: Dietary Supplement: Ketocal 2.5:1

INTERVENTIONS:
Dietary Supplement: Ketocal 2.5:1 — A ketogenic feed for the dietary management of intractable epilepsy is given over a period of four weeks, after a control period of 4 weeks. The amount of the feed given is determined by the Dietitian and/or Doctor responsible for the patient's care (at least one carton per day).

SUMMARY:
An evaluation of the tolerance, compliance, acceptability and safety of a nutritionally complete liquid feed for use as part of the ketogenic diet (KD) in children 8+ years, adolescents and adults with intractable epilepsy or other disorders where the KD is indicated.

DETAILED DESCRIPTION:
An evaluation of the tolerance, compliance, acceptability and safety of a nutritionally complete liquid feed for use as part of the ketogenic diet (KD) in children 8+ years, adolescents and adults with intractable epilepsy or other disorders where the KD is indicated.

Study is conducted over 59 days:

3 day baseline period - Patient continues on whatever dietary regimen they were on before joining the study (this may be a ketogenic diet for existing patients).

28 day control period - Patient begins ketogenic diet (if they are not already on one), and continues this for 28 days WITHOUT the study product. Patients already on a ketogenic diet continue this as normal.

28 day intervention period - A set amount of the study product is incorporated into the patient's ketogenic diet.

Data is captured by the HCP in the case report form at baseline, mid study and end of intervention, and by the patient daily throughout in a patient questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 8 years of age or older
* Diagnosed with intractable epilepsy or another disorder where the KD is indicated
* Motivated to follow the KD for at least the duration of the trial period
* Either currently on a KD, or referred to start a KD
* Likely to benefit from Ketocal 2.5:1
* Written informed consent from patient and/or parent/carer, or completed consultee declaration form
* Willing to take finger prick blood samples to measure ketone levels

Exclusion Criteria:

* Being pregnant or planning pregnancy
* Requiring parenteral nutrition
* Major hepatic or renal dysfunction
* Participation in other clinical intervention studies within 1 month prior to entry of this study
* Allergy to any of the study product ingredients
* Investigator concern around willingness/ability of patient or parent/carer to comply with protocol requirements
* Any contraindications for the use of the ketogenic diet
* Significantly underweight (Body Mass Index <18.5)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal tolerance | Throughout study (59 days)
  GI tolerance will be recorded throughout the study via standardised questionaire

SECONDARY OUTCOMES:
Compliance with feed prescription | Throughout intervention period (28 days)
  Compliance with the study product will be assessed daily throughout the study intervention period by recording how much feed was consumed in mls and comparing this to the amount patients have been prescribed by their Dietitian.
Acceptability and Ease of Use | Measured on day 28 to represent 4 week baseline period, and also measured on day 59 (reflecting 4 week intervention period)
  Acceptability and ease of use will be assessed by questionnaire completed by the parent/carer at the end of the control period (Day 28) for the KD, and at the end of the intervention period (Day 56) for both the diet as a whole and the study product alone.
Adverse events and Seizures | Throughout study (59 days)
  All adverse events and seizures will be monitored throughout the study.
Nutrient intake | Throughout study (59 days)
  Food diaries and 24hr recalls during baseline, control and intervention periods
Height | 59 days (measured at start (day 1), middle (day 31) and end of this period (day 59))
  Height (cm)
Weight | 59 days (measured at start (day 1), middle (day 31) and end of this period (day 59))
  Weight (kg)
Ketone levels | 59 days.
  Blood ketone levels captured via fingerprick blood test 9 days (3 in baseline, 3 in control period and 3 day in the intervention period), twice a day. All other ketone levels alo recorded

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Stratton, PhD, Study Director — Nutricia, University of Southampton.
Locations (9):
- United Kingdom (9):
  - North Bristol NHS Trust, Bristol, Bs105nb
  - University Hospitals Southampton NHS Foundation Trust, Southampton, Hampshire
  - NHS Grampian, Aberdeen
  - Birmingham and Solihull Mental Health NHS Foundation Trust, Birmingham
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Tayside, Dundee
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No